CLINICAL TRIAL: NCT02804295
Title: Collaborative Care From the Emergency Department for Trauma Patients With Prescription Drug Misuse: A Feasibility Study
Brief Title: Collaborative Care From the ED for Trauma Patients With Prescription Drug Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Lauren Whiteside, Acting Assistant Professor, Division of Emergency Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 48977-G
Record Dates: First submitted 2016-06-08; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Substance-Related Disorders
Keywords: Prescription Drug; Misuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Collaborative Care Intervention (Other): All enrolled participants received the collaborative care intervention over 6 months.
  Interventions: Other: Collaborative Care Intervention

INTERVENTIONS:
Other: Collaborative Care Intervention — All eligible subjects that meet the eligibility requirements for approach and consent and have a positive screen for PDM will complete a baseline survey and will be enrolled into the intervention condition. This is an open trial and thus all consenting eligible subjects will receive the intervention.

SUMMARY:
Injured trauma patients in the Emergency Department (ED) may be a particularly important group to target for screening and intervention for prescription drug misuse (PDM). These patients have high rates of psychiatric and substance use co-morbidity and pain management for their injuries (e.g. broken bones, burns) will often require prescribed opioid pain medications and other controlled substances. To date, there are no effective ED-based interventions for PDM. Collaborative Care is a longitudinal model of care that combines multiple elements for patients with complex medical comorbidities. This model holds promise as an intervention strategy for injured patients in the ED that are at risk for prescription drug misuses. Collaborative Care from the ED is innovative and requires developing follow up procedures on a population that has previously been difficult to follow and may have previously avoided consistent health care delivery. The primary objective of this study was to determine the feasibility of initiating a collaborative care intervention for injured ED patients with PDM by enrolling patients into an open trial of this intervention. A secondary objective was to determine if PDM decreases over time after enrollment and developing successful follow-up procedures to deliver longitudinal care.

DETAILED DESCRIPTION:
The investigators will be conducting an open pilot trial of a collaborative care intervention for patients in the Emergency Department (ED) with trauma and prescription drug misuse. Since this is an open trial, all enrolled participants will receive the intervention.

Pre Screen: Prior to approach, the Research Assistant (RA) will review the electronic medical record (EMR) in the ED to first identify patients presenting for an injury and then to determine if they are at risk for prescription drug misuse. The manual chart review information will be entered by the RA into an Excel spreadsheet or equivalent. This process allows the team to identify patients who are at high risk for prescription drug misuse prior to approach.

Approach and Consent: Next, the RA will go to the Emergency Department (ED) or inpatient ward and describe the study to the patient. Informed consent will be obtained from those patients who agree to participate in the protocol.

Eligibility Screening: After consent and enrollment, the RA will provide each consenting subject with a tablet computer so they can self- administer the screening assessment. If the subject requires assistance, the RA can administer the screening assessment. This will include some basic demographic items and a validated survey developed by the National Institute on Drug Abuse (NIDA). Subjects will screen into the study if they have a score of greater than 1 on this validated survey, which indicates having risk for prescription drug misuse. Next, subjects will answer questions regarding contact information including phone number, email and address and travel plans. Since the intervention phase for this study requires multiple contacts and longitudinal engagement, this information is important to inform enrollment. The administration of this stage of screening will take approximately 10-15 minutes. As one of the aims for this study is refining follow-up procedures, every participant must have plans to a) be in the local area for six months (e.g. no long-term travel plans or plans to relocate) b) have at least two contacts and c) have a phone number.

All eligible subjects that meet the eligibility requirements documented above will complete a baseline survey using a tablet computer and will be enrolled into the intervention condition. This is an open trial and thus all consenting eligible subjects will receive the intervention.

Collaborative Care Intervention: Subjects that are eligible for the intervention after screening will be visited by a study care manager at the bedside in the hospital. This care manager will use motivational interviewing techniques to elicit and target for improvement each subject's unique constellation of concerns and needs. The care manager will also ask about treatment preferences and will schedule ongoing times to meet/call the subject during the initial days and weeks post-injury. The care manager will give the subject the study team's 24-hour contact number and encourage calls for spontaneous questions, needs, and concerns. These subjects will be given a choice of treatment options and the care manager will share information and deliberate medical treatment decisions with each subject. Together the care manager and subject will develop a treatment plan informed by each subject's injury and medical needs, substance abuse needs, prescription medication needs and concerns. The collaborative care intervention will be comprised of the following elements based on participant's need:

1. Medication Management: This element of the intervention will focus on appropriate medication guidelines for prescription opioids, and patient comorbidities as well as providing guideline adherence recommendations for opioid prescribing in acute and primary care settings.
2. Care coordination and linkage: Intervention team members will work collaboratively with acute and primary care providers in an effort to coordinate care longitudinally through outpatient follow-up. The care manager will meet subjects at their outpatient appointments whenever possible. The care manager will also attempt to establish primary care linkages for each subject. Stepped, higher intensity care linkages will be available for subjects with severe mental health needs or substance abuse needs.
3. Care management:

Care manager supervision: After the initial evaluation, the care manager will discuss each participant and their needs with study PI and team. As indicated, the PI and/or the care manager will be in contact with study participants via phone after team meetings to monitor side effects of new medications or for adjustments to the recommended pharmacotherapy plan. The care manager will receive standard clinical supervision delivered by study members.

Follow-up Assessments: Each participant will be contacted to complete a follow-up assessment at 1-month, 3-months and 6-months after their hospital visit for injury. The follow-up assessment will be completed in person, over the phone or via internet using the method preferred by the participant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-65 years old) presenting to Harborview Medical Center in Seattle, Washington with an injury from 02/2015 to 09/2015 were screened for eligibility based on historical codes in the electronic medical record (EMR) that increase their risk for prescription drug misuse. The items pulled from electronic medical charts for a pre-screen include: History of opioid, sedative or stimulant abuse or dependence, history of opioid overdose, current opioid prescriptions, co-occurring prescriptions for opioids and sedatives, previous ED visit at Harborview Medical Center (HMC) attributable to substance use, number of ED visits in the past year. Possible participants who met this eligibility criteria were approached by the research assistant. Consented patients completed a screening assessment for PDM based on NIDA m-ASSIST for prescription opioids, sedatives and stimulants and select questions from the Current Opioid Misuse Measure. Participants with a positive screen for PDM were enrolled in the 'Prescription Collaborative Care (RxCC)' intervention.

Exclusion Criteria:

* Participants were excluded if they were incarcerated or under arrest, required active resuscitation in the ED or other clinical area at the time of RA approach, had a diagnosis of cancer or are receiving palliative or hospice care, were in the ED or hospital for a primary psychiatric emergency such as suicidal ideation or attempt, lived beyond a 50 mile radius of HMC, or did not have reliable contact information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Establishing the Feasibility of a Collaborative Care Intervention by Measuring the Rate of Patient Consent | This outcome was measured during active recruitment of patients in the ED until recruitment completion, which lasted 5 months.
  The primary outcome of intervention feasibility was assessed by measuring the rate of eligible patients that consented and enrolled in the intervention upon approach by the research assistant.
Establishing the Acceptability of a Collaborative Care Intervention by Measuring the Proportion of Enrolled Patients that Completed the Intervention in the ED | This outcome was measured during active recruitment of patients in the ED until recruitment completion, which lasted 5 months.
  The primary outcome of intervention acceptability was assessed by measuring the proportion of consented patients that completed the collaborative care intervention in the ED with members of the intervention team.

SECONDARY OUTCOMES:
Self-Reported Patient Satisfaction Using the Client Satisfaction Questionnaire-8 (CSQ-8) | Patient satisfaction was measured upon completion of the intervention for each patient, after the patient's 6-month follow-up assessment. Measurement for this outcome lasted approximately 6 months.
  This outcome measures self-reported patient satisfaction with the collaborative care intervention as assessed by the Client Satisfaction Questionnaire-8 (CSQ-8).
Self-Reported Health Care Utilization of Enrolled Patients Throughout the Study Duration | Patients self-reported their health care utilization at the time of enrollment and at 1-, 3-, and 6-month follow-up assessments. This was assessed through study completion (approximately 1 year).
  Patients self-reported their health care utilization (including ED utilization, visits to primary care doctors, specialists, etc.) at time of enrollment (health care utilization for the past 6 months) and at 1-, 3-, and 6-month follow-up assessments (health care utilization since last assessment).
Self-Reported Substance Use of Enrolled Patients as Assessed by the NIDA Modified-Alcohol, Smoking, and Substance Involvement Screening Test (NM-ASSIST) | Patients self-reported their substance use at the time of enrollment and at 1-, 3-, and 6-month follow-up assessments. This was assessed through study completion (approximately 1 year).
  Patients self-reported their substance use using the NM-ASSIST measure at time of enrollment (reported substance use for the past 6 months) and at 1-, 3-, and 6-month follow-up assessments (reported substance use since last assessment).
Follow-up Retention Rates | Follow-up rates for enrolled patients at 1-, 3-, and 6-months post enrollment were measured throughout the duration of the study through study completion, which lasted approximately one year.
  Follow-up retention rates of enrolled patients (i.e. patients that complete follow-up assessments at 1-, 3-, and 6-months post enrollment) are measured for each follow-up assessment time period (1-, 3-, and 6-months post enrollment). These follow-up assessments began 1-month after the first subject was recruited and continued for up to 6 months after the recruitment of the last subject.

IPD SHARING:
Plan to Share IPD: No